CLINICAL TRIAL: NCT06041074
Title: The Clinical Characteristics of Adenoid Vegetations in Adult Patients
Brief Title: Adenoid Vegetations in Adult Patients
Status: Completed | Type: Observational
Sponsor: Varazdin General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1968
Record Dates: First submitted 2023-09-05; First posted 2023-09-18 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-09

CONDITIONS: Adenoid Vegetation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults: Patients with adenoid vegetations, 14 years old and older
- Children: Patients with adenoid vegetations, 13 years old and younger

SUMMARY:
In this observational cross-sectional study " the clinical characteristics of adenoid vegetations in adulthood will be investigated.

DETAILED DESCRIPTION:
Adenoid vegetations typically appear in childhood and are well described in this population. However, in adulthood, adenoid vegetations appear rarely and their characteristics have not been described.

The clinical characteristics of adenoid vegetations in adulthood will be investigated, and compared with clinical characteristics of adenoid vegetations in childhood.

ELIGIBILITY:
Inclusion Criteria:

* patient with adenoid vegetations

Exclusion Criteria:

* other concomitant otorhinolaryngological diagnoses
* hypertrophy of the tonsils
* oropharyngeal carcinomas
* chronic sinuitis
* allergic rhinitis

Ages: 1 Year to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult group: All patients aged 14 and more treated for adenoid vegetations in Varazdin General Hospital from 1 January 2013 to 31 December 2019
  Children group: All patients aged 13 and less treated for adenoid vegetations in Varazdin General Hospital from 1 January 2019 to 31 December 2019
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Symptoms | 2 months
  The leading symptom (patient's main complaint, the reason for seeing the doctor) will we recorded for each participant

SECONDARY OUTCOMES:
Duration of symptoms | 2 months
  The duration of leading symptom (in months) will be recorded for each participant
OTS (otoscopic) | 2 months
  The otoscopic findings will be recorded in both groups
RNS (rhinoscopic) | 2 months
  The rhinoscopic findings will be recorded in both groups
OFS (oropharyngoscopic) | 2 months
  The oropharyngoscopic findings will be recorded in both groups
PRNS (post-rhynoscopic) | 2 months
  The post-rhynoscopic findings will be recorded in both groups
Referring physician | 2 months
  The physician (primary or secondary level) who referred the patient to ENT (Ear Nose and Throat doctor) will be recorded in both groups
PHD ( pathohistological findings) | 2 months
  The pathohistological findings will be recorded in both groups
Surgery | 2 months
  The type of surgery will be recorded in both groups
Outcome | 2 months
  The outcome (the relief of the leading symptom) will be recorded in both groups
Recurrence | 2 months
  The recurrence will be recorded in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Drazen Shejbal, Principal Investigator — Varazdin General Hospital, Varazdin, Croatia
Locations (1):
- Varazdin General Hospital, Varaždin, Croatia